CLINICAL TRIAL: NCT01020136
Title: A Phase 1 Bioequivalence Study To Compare The Plasma Pharmacokinetics Of AG-013736 Polymorph Form IV Versus Market-Image Polymorph Form XLI Tablets In Healthy Volunteers Under Fed Conditions
Brief Title: A Bioequivalence Study Of AG-013736 Tablets Under Fed Conditions In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A4061063
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2010-04-22 (Estimated); Status verified 2010-04

CONDITIONS: Healthy Volunteer
Keywords: Bioequivalence Pharmacokinetics
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (BABA) (Experimental): Treatment A: 5-mg Form IV tablet; Treatment B: 5-mg Form XLI tablets Subjects in this sequence will participate in 4 periods in the following order: B -> A -> B -> A
  Interventions: Drug: AG-013736
- Sequence 2 (ABAB) (Experimental): Treatment A: 5-mg Form IV tablet; Treatment B: 5-mg Form XLI tablets Subjects in this sequence will participate in 4 periods in the following order: A -> B-> A -> B
  Interventions: Drug: AG-013736

INTERVENTIONS:
Drug: AG-013736 — single oral dose 5-mg tablet (Form IV for Treatment A and Form XLI for Treatment B under fed conditions)
  Arms: Sequence 1 (BABA)
Drug: AG-013736 — single oral dose 5-mg tablet (Form IV for Treatment A and Form XLI for Treatment B under fed conditions)
  Arms: Sequence 2 (ABAB)

SUMMARY:
The purpose is to show that 5 mg Form IV tablet of AG-013736 produces similar drug concentrations in plasma compared to 5 mg Form XLI tablet of AG-013736 after oral dosing under fed conditions.

DETAILED DESCRIPTION:
To establish bioequivalence between Form IV and Form XLI of AG-013736 tablets

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 47 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead electrocardiogram (ECG) and clinical laboratory tests)
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs)
* An informed consent document signed and dated by the subject or a legally acceptable representative

Exclusion Criteria:

* Evidence of significant disease of the blood, kidney, endocrine system, lungs, gastrointestinal, heart, liver, psychiatric, neurologic, or allergic (including drug allergies, but excluding season allergies)
* Use of tobacco- or nicotine- containing products (or a positive urine cotinine test).
* Pregnant or nursing females and females of childbearing potential including those with tubal ligation

Ages: 21 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To establish the bioequivalence of test 5 mg market-image tablets of AG-013736 polymorph Form XLI to reference 5 mg tablets of AG- 013736 polymorph Form IV under fed conditions. | 3 days per period

SECONDARY OUTCOMES:
To assess the safety and tolerability of single dose AG-013736 when administered as polymorph Forms XLI and IV in healthy volunteer | 3 days per period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061063&StudyName=A%20Bioequivalence%20Study%20Of%20AG-013736%20Tablets%20Under%20Fed%20Conditions%20In%20Healthy%20Volunteers